CLINICAL TRIAL: NCT02708082
Title: Glaucoma HFA / OCT Specificity Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Carl Zeiss Meditec, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: COMBO-2015-1
Record Dates: First submitted 2016-02-24; First posted 2016-03-15 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Glaucoma: Early, moderate or advanced glaucoma, glaucoma suspects or pre-perimetric glaucoma will perform OCT scanning and HFA perimetry
  Interventions: Device: OCT scanning and HFA perimetry

INTERVENTIONS:
Device: OCT scanning and HFA perimetry — Imaging of the optic nerve and nerve fiber layer / measurement of visual field

SUMMARY:
Study consists of five visits over a one to three month time period.

DETAILED DESCRIPTION:
Each visit consists of optical coherence tomography (OCT) scanning (4 scans ) and two HFA (Humphrey Field Analyzer) visual fields of the study eye only.

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females 40 to 80 years old
* Able and willing to attend the required study visits
* Able and willing to provide consent and follow study instructions in English
* A diagnosis by the Principal Investigator or co-investigator of glaucoma, pre-perimetric glaucoma or glaucoma suspect
* Subjects must have experience in threshold automated perimetry, having performed a previous SITA (Swedish Interactive Thresholding Algorithm) threshold test within one year of enrolling to the study
* Ability to fixate that allows obtaining acceptable visual fields and OCT scans in the study eye

Exclusion Criteria:

* • Best-corrected visual acuity less than 20/40 (study eye only) on a Snellen chart or on a Snellen equivalent acuity chart

  * Spherical refraction outside -12.00 to +5.00 diopters (D) or cylinder correction outside 3.00 D (study eye only)
  * Amblyopia (either eye)
  * Narrow irido-corneal angles or a diagnosis of narrow angle glaucoma
  * Previous or current eye disease in the study eye, serious eye trauma or intraocular surgery (except cataracts with lens implants), or the presence of ocular findings that could affect the visual field, other than glaucoma
  * Cataract surgery in the study eye within six (6) months of first visit
  * Dx of any optic neuropathy other than glaucoma
  * Vitreoretinal traction or epiretinal membrane in the study eye
  * Diagnosis or history of any systemic disease / condition / treatment which is likely to affect the visual field outcome in the Study Eye other than glaucoma
  * History of diabetes, leukemia, AIDS, uncontrolled systemic high blood pressure, dementia or multiple sclerosis
  * Any disease that is likely to progress within the 3 month time period that might have visual field implications
  * A life threatening or debilitating disease
  * Participation in any study involving a non-FDA approved investigational drug (IND) within the past month, or ongoing participation in a study with a non-FDA approved or cleared investigational device (IDE)
  * Concomitant use of hydrochloroquine and/or chloroquine

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult males or females 40 to 80 years old with diagnosis of glaucoma, pre-perimetric glaucoma or glaucoma suspect
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-08 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Retinal nerve fiber layer average thickness | less than 3 months
  Specificity comparison of results from the five visits will be made. Analysis of variance will be used to determine repeatability and reproducibility - results in microns.

SECONDARY OUTCOMES:
Neuroretinal rim thickness | less than 3 months
  Specificity comparison of results from the five visits will be made. Analysis of variance will be used to determine repeatability and reproducibility - results in millimeters squared.
Mean deviation of visual field | less than 3 months
  Specificity comparison of results from the five visits will be made. Analysis of variance will be used to determine repeatability and reproducibility - results in decibels.
Pattern standard deviation of the visual field | less than 3 months
  Specificity comparison of results from the five visits will be made. Analysis of variance will be used to determine repeatability and reproducibility - results in decibels.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Callan, Study Director — Carl Zeiss Meditec, Inc.
Locations (1):
- Carl Zeiss Meditec, Inc., Dublin, California, United States

IPD SHARING:
Plan to Share IPD: No